CLINICAL TRIAL: NCT06100289
Title: An Open-Label, Phase 3 Study to Evaluate the Pharmacokinetics, Safety, and Immunogenicity of Vedolizumab Subcutaneous in Pediatric Subjects With Moderately to Severely Active Ulcerative Colitis or Crohn's Disease Who Achieved Clinical Response Following Open-Label Vedolizumab Intravenous Therapy
Brief Title: A Study of Vedolizumab in Children and Teenagers With Ulcerative Colitis or Crohn's Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VedolizumabSC-3003; 2023-503188-40-00 (EU CTIS Number: Abbreviated EU CT Number); jRCT2071240072 (Registry Identifier: jRCT)
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Induction Period: Participants ≥30 kg, Vedolizumab (High Dose) IV (Experimental): Participants weighing ≥30 kg will receive vedolizumab (High Dose) IV infusion, at Day 1, Weeks 2 and 6 in the Induction Period.
  Interventions: Drug: Vedolizumab IV
- Induction Period: Participants >15 to <30 kg, Vedolizumab (Medium Dose) IV (Experimental): Participants weighing >15 to <30 kg will receive vedolizumab (Medium Dose), IV infusion, at Day 1, Weeks 2 and 6 in the Induction Period.
  Interventions: Drug: Vedolizumab IV
- Induction Period: Participants ≥10 to ≤15 kg, Vedolizumab (Low Dose) IV (Experimental): Participants weighing ≥10 to ≤15 kg will receive vedolizumab (Low Dose), IV infusion, at Day 1, Weeks 2 and 6 in the Induction Period.
  Interventions: Drug: Vedolizumab IV
- Maintenance Period: Participants ≥30 kg, Vedolizumab 108 mg SC Q2W (Experimental): Participants with clinical response at Week 14 weighing ≥30 kg will receive vedolizumab 108 mg, SC injection, Q2W from Week 14 to Week 32 in the Maintenance Period.
  Interventions: Drug: Vedolizumab SC
- Maintenance Period: Participants ≥10 to <30 kg, Vedolizumab 108 mg SC Q4W (Experimental): Participants with clinical response at Week 14 weighing ≥10 to <30 kg will receive vedolizumab 108 mg, SC injection, Q4W from Week 14 to Week 30 in the Maintenance Period.
  Interventions: Drug: Vedolizumab SC

INTERVENTIONS:
Drug: Vedolizumab IV — Vedolizumab IV injection.
  Other Names: ENTYVIO; KYNTELES; MLN0002
  Arms: Induction Period: Participants >15 to <30 kg, Vedolizumab (Medium Dose) IV; Induction Period: Participants ≥10 to ≤15 kg, Vedolizumab (Low Dose) IV; Induction Period: Participants ≥30 kg, Vedolizumab (High Dose) IV
Drug: Vedolizumab SC — Vedolizumab SC injection.
  Other Names: MLN0002SC
  Arms: Maintenance Period: Participants ≥10 to <30 kg, Vedolizumab 108 mg SC Q4W; Maintenance Period: Participants ≥30 kg, Vedolizumab 108 mg SC Q2W

SUMMARY:
The main aim of this study is to learn how the body of a child or teenager with moderately to severely active ulcerative colitis (UC) or Crohn's disease (CD) processes vedolizumab (pharmacokinetics) given just under the skin subcutaneously (SC).

The participants will be treated with vedolizumab for up to 34 weeks.

During the study, participants will visit their study clinic several times.

DETAILED DESCRIPTION:
The drug being tested in this study is vedolizumab. Vedolizumab is being tested to treat pediatric participants with moderate to severe active UC or CD who achieved clinical response following open-label vedolizumab intravenous (IV) therapy. The study will look at the pharmacokinetics, safety, and immunogenicity of vedolizumab.

The study will enroll approximately 70 patients. During the Induction Period participants will receive 3 doses of vedolizumab IV infusion at Day 1, Week 2, and Week 6 based on their weight at Baseline as:

* Participants ≥30 kilograms (kg), Vedolizumab (High Dose)
* Participants >15 to <30 kg, Vedolizumab (Medium Dose)
* Participants ≥10 to ≤15 kg, Vedolizumab (Low Dose)

At Week 14, participants who achieve clinical response will be assigned to one of the following groups, stratified by weight to receive vedolizumab 108 mg SC injection during the 20-week Maintenance Period:

* Participants ≥30 kg, Vedolizumab 108 mg once every 2 weeks (Q2W)
* Participants ≥10 to <30 kg, Vedolizumab 108 mg once every 4 weeks (Q4W)

This multi-center trial will be conducted globally. After the Week 34 end of treatment (EOT) visit assessments have been completed, participants may be eligible to receive continued treatment with vedolizumab SC in an extension study, whereas participants who do not qualify to receive continued treatment in the extension study or participants who discontinue from the study for any reason will complete the EOT visit, and the follow-up safety visit (18 weeks after last dose).

ELIGIBILITY:
Inclusion Criteria:

1. The participant weighs ≥10 kg at the time of screening and enrollment into the study.
2. Participants with UC or CD diagnosed at least 1 month before screening. Participants with moderately to severely active disease defined as:

   * Participants with UC: a modified Mayo score of 5 to 9 (sum of Mayo endoscopic subscore, stool frequency subscore, and rectal bleeding subscore) with a Mayo endoscopic subscore of ≥2 (with the presence of mucosal friability excluding an endoscopic subscore of 1 and mandating a score of at least 2). (The results of screening endoscopy should be applied.)
   * Participants with CD: a pediatric Crohn's disease activity index (PCDAI) >30 and a simple endoscopic score for Crohn's disease (SES-CD) >6 (or an SES-CD ≥4 if disease is confined to terminal ileum) at screening endoscopy.
3. Participants who have failed, lost response to, or been intolerant to treatment with at least 1 of the following agents: corticosteroids, immunomodulators (for example, azathioprine [AZA], 6-mercaptopurine [6-MP], methotrexate [MTX]), and/or tumor necrosis factor (TNF)-α antagonist therapy (for example, infliximab, adalimumab).
4. Participants with evidence of UC extending proximal to the rectum (that is, not limited to proctitis), at a minimum.
5. Participants with extensive colitis or pancolitis of >8 years' duration or left-sided colitis of >12 years' duration must have documented evidence of a negative surveillance colonoscopy within 12 months before screening.
6. Participants with vaccinations that are up-to-date based on the countrywide accepted schedule of childhood vaccines.

Exclusion Criteria:

1. Participants who have had previous exposure to approved or investigational anti-integrins, including but not limited to, natalizumab, efalizumab, etrolizumab, or abrilumab (AMG 181); or mucosal addressin cell adhesion molecule-1 (MAdCAM-1) antagonists (ontamalimab), or rituximab.
2. Participants who have had prior exposure to vedolizumab.
3. Participants with hypersensitivity or allergies to vedolizumab or any of its excipients.
4. Participants with active cerebral/meningeal disease, signs/symptoms or history of progressive multifocal leukoencephalopathy (PML) or any other major neurological disorders.
5. The participant has received any live vaccinations within 30 days before first dose of study drug.
6. Participants who currently require surgical intervention or are anticipated to require surgical intervention for UC or CD during this study.
7. Participants who have had subtotal or total colectomy or have a jejunostomy, ileostomy, colostomy, ileo-anal pouch, known fixed stenosis of the intestine, short bowel syndrome, or >3 small intestine resections.
8. Participants with a current diagnosis of indeterminate colitis.
9. Participants with clinical features suggesting monogenic very early-onset inflammatory bowel disease (IBD).
10. Participants with active or latent tuberculosis (TB).
11. Participants with evidence of positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Hepatitis B virus (HBV) immune subjects (that is, HBsAg negative and hepatitis B surface antibody [anti-HBs]-positive) may, however, be included.
12. The participant has any identified congenital or acquired immunodeficiency (for example, common variable immunodeficiency, human immunodeficiency virus [HIV] infection, organ transplantation).
13. Participants with positive stool studies for ova and/or parasites or stool culture at screening visit.
14. Participants with positive Clostridioides difficile (C difficile) stool test at screening visit.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Ctrough,ss: Steady-state Median Observed Plasma Concentration at the End of a Dosing Interval for Vedolizumab at Week 34 | Predose at Week 34
Cavg,ss: Average Serum Concentration at Steady-state for Vedolizumab at Week 34 | Multiple time points prior to Week 34; pre-dose at Week 34

SECONDARY OUTCOMES:
Percentage of Participants with Positive Antivedolizumab Antibody (AVA) | Baseline up to 18 weeks after last dose of study drug (up to Week 50)
Percentage of Participants with Positive Neutralizing AVA | Baseline up to 18 weeks after last dose of study drug (up to Week 50)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (57):
- United States (11):
  - VVCRD Clinical Research, Garden Grove, California
  - Loma Linda University School of Medicine, Loma Linda, California
  - Children's Hospital Of Orange County, Orange, California
  - Stanford Children's Health, Palo Alto, California
  - Advocate Children's Hospital, Park Ridge, Illinois
  - Children's Hospital of Michigan, Detroit, Michigan
  - Atlantic Health System, Morristown, New Jersey
  - New York Presbyterian Hospital, Weill Cornell Medical College, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina, North Charleston, South Carolina
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Centre Hospitalier Chretien MontLegia, Liège
- Bulgaria (2):
  - University Hospital "Saint George", Plovdiv
  - Specialized Hospital for Active Treatment of Children Diseases "Prof. Dr. Ivan Mitev" EAD, Sofia
- Denmark (2):
  - Hvidovre University Hospital, Hvidovre, Capital Region
  - H.C Andersens Hospital, Odense
- Childrens Health Ireland, Dublin, Ireland
- Italy (4):
  - Azienda Ospedaliera Universitaria Gaetano Martino Messina, Messina
  - V. Buzzi Hospital, Milan
  - Unita Operativa Complessa Di Pediatria Medica, Pescara
  - IRCCS Ospedale Pediatrico Bambino Gesu, Rome
- Japan (3):
  - Kurume University Hospital, Kurume, Fukuoka
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - National Center for Child Health and Development (NCCHD), Setagaya-Ku, Tokyo
- Radboud University Medical Center, Nijmegen, Netherlands
- Poland (5):
  - Instytut Pomnik - Centrum Zdrowia Dziecka, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Dzieciecy W Krakowie, Krakow
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Medical Network Sp. Z.o.o. WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - SPSK Nr 1 im. Prof. S. Szyszko SUM w Katowicach, Zabrze
- Portugal (3):
  - Hospital Pediatrico - Unidade Local de Saude de Coimbra, Coimbra
  - Hospital St Maria- Centro Hospitalar de Lisboa, Norte EPE, Lisbon
  - Centro Materno Infantil do Norte - Unidade Local de Saude de Santo Antonio, Porto
- Romania (3):
  - "Emergency County Clinical Hospital ""Pius Brinzeu""", Timișoara, Timiș County
  - Dr Victor Gomoiu Clinical Children Hospital, Bucharest
  - Spitalul Clinic de Urgenta Pentru Copii ,,Grigore Alexandrescu,, Bucharest
- Serbia (3):
  - University Children's Hospital, Belgrade
  - Mother and child helath care Institute of Serbia dr Vukan Cupic, Belgrade
  - Institute for Childand YouthHealth Care of Vojvodina, Novi Sad
- South Korea (4):
  - Kyungpook National University Chilgok Hospital (KNUCH), Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Complejo Hospitalario Universitario de Ferrol, Ferrol
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital U. Virgen Macarena, Seville
  - Hospital Univesritario y Politecnico La Fe. Av Fernando abril Martorell106. Valencia 46026. Spain, Valencia
- Switzerland (3):
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Inselspital, Universitatsspital Bern, Kinderklinik, Julie-von-Jenner-Haus, Bern
  - Universitats-Kinderspital, Zurich
- Taiwan (3):
  - National Taiwan University Children's Hospital, Taipei, Zhongzheng Dist
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
- Turkey (Türkiye) (3):
  - Koc University Hospital, Istanbul, Zeytinburnu
  - Istanbul University, Istanbul Medical Faculty, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/a010ca2923444630?idFilter=%5B%22VedolizumabSC-3003%22%5D